CLINICAL TRIAL: NCT06606834
Title: Assessment of the Uterus Using Ultrasonographic Elastography in Women with Dysmenorrhea
Status: Not yet recruiting | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Bilge Pinar Keskinsoy, MD, Ufuk University
Other Study IDs: 24.06.11.02/01
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Sonoelastography
MeSH Terms: conditions — Dysmenorrhea | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: sonoelastography — Elasticity is defined as the ability of an organ or tissue to return to its original shape after being deformed by an applied force or stress. Based on this principle, sonoelastography is a technique used to assess the elasticity of tissues and organs during ultrasonography. This assessment allows measurement of changes in stiffness of soft tissues following physiological or pathological processes.

SUMMARY:
The aim of this study is to perform sonoelastographic assessment of the uterus in patients diagnosed with primary dysmenorrhea and to compare these measurements with sonoelastographic evaluations of the uteri in asymptomatic individuals. This will enable, for the first time, the demonstration of whether the elasticity of the myometrial tissue contributes to the etiology of primary dysmenorrhea.

Secondary Objectives: To determine whether there is a correlation between the severity of primary dysmenorrhea and ultrasonographic markers.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40 years.
2. Women with primary dysmenorrhea who are willing to participate in the study.
3. Women without primary or secondary dysmenorrhea who agree to participate as a control group.

Exclusion Criteria:

1. Women with secondary dysmenorrhea.
2. Patients with underlying uterine or adnexal pathologies (e.g., endometrial polyps, adenomyosis, uterine fibroids, adnexal masses, ovarian pathologies and cysts) identified via ultrasonography.
3. Individuals with a history of uterine surgery.
4. Individuals with a history of pelvic surgery.
5. Individuals who have delivered via normal spontaneous vaginal delivery or cesarean section.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: dysmenorrhea patient group
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
SWE Tecnique | 1 year
  The SWE technique, available in the ultrasound device software, will be used with no additional cost to the patient or institution. With SWE, at least 3 different measurements will be taken from the closest myometrial layer in both axial and sagittal planes, and both speed and elasticity values will be recorded as minimum, maximum, and mean values. The speed of shear waves increases as tissue hardness increases, therefore there is a direct proportion between tissue elasticity and velocity. The elasticity of the tissue is measured with the formula G(tissue elasticity)= ρ(tissue density)c²(shear wave velocity), also called shear modulus. While tissue elasticity is obtained in Kpa, the unit of tissue density is kg/m³ and the shear wave velocity is expressed in m/sn.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided